CLINICAL TRIAL: NCT02989246
Title: Effort of Breathing Guided Ventilator Management for Children Using Pressure Rate Product: a Pilot Study
Brief Title: Effort of Breathing Guided Ventilator Protocol
Acronym: EOBvent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Robinder Khemani, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-14-00473
Record Dates: First submitted 2016-12-06; First posted 2016-12-12 (Estimated); Results first posted 2021-10-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Ventilators, Mechanical; Work of Breathing
Keywords: pediatrics; ventilator weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Ventilator management using the proposed protocol in both acute and weaning phases. Patients will be managed according the the Ventilator protocol using the esophageal catheter for the weaning phase
  Interventions: Other: Ventilator protocol; Device: Esophageal Catheter

INTERVENTIONS:
Other: Ventilator protocol — Open loop ventilator management by a computer based protocol
Device: Esophageal Catheter — Esophageal manometry measurements of patient effort of breathing will be used to guide the protocol recommendations

SUMMARY:
This pilot study tests the feasibility of using a computerized ventilator management protocol seeking to encourage lung protective ventilation during the acute phase of ventilation, and esophageal manometry based titration of ventilator settings during the weaning phase of ventilation, for children with acute respiratory failure. The investigators hypothesize that such an approach will reduce time on mechanical ventilation, largely by preserving diaphragm muscle function.

DETAILED DESCRIPTION:
Objectives: This pilot study will help refine a computer based ventilator management protocol which will be used in both acute and weaning phases of ventilation for children with acute respiratory failure. The acute phase protocol is an adaptation of the Acute Respiratory Distress Syndrome Network protocol for pediatrics, and the weaning phase involves an esophageal manometry guided weaning protocol based on effort of breathing. The investigators seek to test the safety and feasibility of the protocol recommendations and the software system , and help determine the potential effect size of the intervention to determine feasibility of a randomized controlled trial. They also seek to determine the feasibility and reproducibility of serial diaphragm ultrasound measurements on mechanically ventilated children.

Study Population: All children intubated and mechanically ventilated in the Children's Hospital Los Angeles Pediatric ICU with an anticipated length of intubation > 48 hours will be eligible, with some exclusion criteria based on ability to perform the measurements.

Study methodology: After consent, an esophageal catheter will be placed. A software management tool for ventilator management will be placed at the bedside for each enrolled patient, and recommendations regarding changing ventilator support will be provided to the clinicians every several hours during both acute and weaning phases. When ventilator support is below a threshold, recommendations will be made to perform spontaneous breathing trials. The clinicians will ultimately decide whether to accept or reject the recommendations, and will evaluate the patient before each potential change to the ventilator. The acceptance or rejection of recommendations will be tracked, and used to refine the intervention. Daily diaphragm ultrasound measurements will also be obtained to monitor diaphragm thickness and contractile activity.

Follow up: Clinical outcomes will be followed while in the ICU including re-intubation, medications administered, and ICU length of stay. No follow up after ICU discharge is planned.

Analysis plans: Data will be used to refine the intervention, test the acceptability of protocol recommendations to bedside providers, and determine sample size estimates for a follow up randomized controlled trial. These analyses will be descriptive. A pilot of 40 patients is anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated patients in the Children's Hospital Los Angeles Pediatric ICU
* Anticipated length of intubation > 48 hours.
* The primary attending physician approves use of the protocol on the patient.

Exclusion Criteria:

* Corrected gestational age less than 37 weeks
* Contraindications to nasoesophageal catheter placement (nasopharyngeal or esophageal abnormalities) or Respiratory Inductance Plethysmography bands (abdominal wall defects such as omphalocele).
* Significant lower airway obstruction (asthma or bronchiolitis), confirmed by ventilator spirometry

Ages: 37 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02-01; Primary Completion 2017-10-18 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robinder Khemani, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No exclusion of patients prior to assignment to the intervention.
Groups:
- Intervention Arm: Ventilator management using the proposed protocol in both acute and weaning phases. Patients were managed according the the Ventilator protocol using the esophageal catheter
  Ventilator protocol: Open loop ventilator management by a computer based protocol
  Esophageal Catheter: Esophageal manometry measurements of patient effort of breathing were used to guide the protocol recommendations
Period: Overall Study
Arm/Group | Intervention Arm
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 32
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 100.7 [30.7 to 150.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Protocol Recommendations Which Are Accepted by the Clinical Provider
Description: The investigators will track the percentage of recommendations which are accepted by providers, as well as the reasons why recommendations were not accepted
Time Frame: With each protocol recommendation, approximately every 4 hours during the course of mechanical ventilation (up to 28 days)
Measure: Mean (95% Confidence Interval); unit: percentage adherant
Arm/Group | Intervention Arm
Number analyzed (Participants) | 32
percentage adherant | 76 [74.8 to 77.9]

ADVERSE EVENTS:
Time Frame: During ICU admission
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 7/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT02989246/Prot_SAP_000.pdf